CLINICAL TRIAL: NCT02689583
Title: A Multi-center Study for Individual Treatment of Helicobacter Pylori Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Peking Union Medical College Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Third Affiliated Hospital of Third Military Medical University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Centers for Disease Control and Prevention, China (Other Government); Academy Military Medical Science, China (Industry)
Responsible Party: Principal Investigator, Youming Li, Director of the Department of Gastroenterology, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FirstZhejiangU YMLi
Record Dates: First submitted 2016-02-01; First posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Gastritis; Gastric Ulcer
Keywords: Helicobacter pylori; Antibiotic resistance; Sequencing; Mechanism; Cause
MeSH Terms: conditions — Gastritis; Stomach Ulcer

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Successful treatment (Experimental): The patients with H. pylori infection have successful treatment based on the results from antibiotic susceptibility testing，CYP2C19 gene polymorphism，drug resistance gene sequencing and 16SrRNA sequencing.
  Interventions: Biological: Antibiotic selection based on the antibiotic susceptibility testing; Genetic: PPI selection based on the CYP2C19 gene polymorphism; Dietary Supplement: Probiotics usage based on the 16SrRNA sequencing
- refractory infection (Experimental): The patients with H. pylori infection have failed treatment based on the results from antibiotic susceptibility testing，CYP2C19 gene polymorphism，drug resistance gene sequencing and 16SrRNA sequencing.
  Interventions: Biological: Antibiotic selection based on the antibiotic susceptibility testing; Genetic: PPI selection based on the CYP2C19 gene polymorphism; Dietary Supplement: Probiotics usage based on the 16SrRNA sequencing

INTERVENTIONS:
Biological: Antibiotic selection based on the antibiotic susceptibility testing — The biological intervention focused on the results from the antibiotic susceptibility testing. All patients should used the their susceptibility antibiotics according to antibiotic susceptibility testing of H. pylori. Considering the safety of drug usage, priority antibiotic selection was as follow: Amoxicillin > Clarithromycin > Levofloxacin >Tetracycline > Furazolidone > Metronidazole.
Genetic: PPI selection based on the CYP2C19 gene polymorphism — PPI selection should based on the CYP2C19 gene polymorphism of patients. Patients have different metabolizers, such as poor metabolizers (PM), extensive metabolizers (EM) and intermediate metabolizer (IM). Different metabolism of patients should select different PPI or different doses of PPI. For IM and PM, in this study, patients selected the standard dose of Omeprazole. For EM, in this study, patients selected the Esomeprazole with increasing doses 50%-100%.
Dietary Supplement: Probiotics usage based on the 16SrRNA sequencing — Different micro-environment in stomach may influence the antibiotic absorption. In this study, some patients could select probiotic as adjuvant therapy according to their micro-environment in stomach by 16SrRNA sequencing.

SUMMARY:
Since the discovery of Helicobacter pylori (H. pylori), many studies have been carried out with the goal of improving H. pylori eradication and therapies have changed from single-antibiotic treatments to the current multi-antibiotic treatments. However, the eradication rate of H. pylori is still less than 80%. The reasons for this low eradication rate are likely to be multi-factorial, including the reduced activity of antimicrobial drugs, poor patient compliance or micro-environment in stomach. In this study, to obtain the higher eradication of H. pylori and discover the different mechanism between the current infection and refractory infection of H. pylori, it is necessary to perform a prevalence survey for eradication of H. pylori based on the results from isolation of H. pylori strains, antibiotic susceptibility testing, CYP2C19 gene polymorphism, drug resistance gene sequencing and 16SrRNA sequencing.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~70 years old, male or female, untreated patients.
2. Symptoms of abdominal pain, bloating, acid reflux, belching, nausea, vomiting, heartburn, chest pain, vomiting, melena, etc.
3. Unused antibiotics, bismuth, H2 receptor antagonists or PPI by nearly 4 weeks 4. 13C-labelled urea breath test positive.

5.Agreed to Helicobacter pylori culture and sensitivity testing taken by endoscopy gastric biopsy specimens,and the result of culture was positive.

6.Agreed to Helicobacter pylori eradication therapy and cooperate with the eradication efficacy follow-up survey.

Exclusion Criteria:

1. Severe heart, liver, kidney dysfunction.
2. Pregnant or lactating women.
3. Complications of bleeding, perforation, pyloric obstruction, cancer.
4. Esophageal,gastrointestinal surgery history.
5. Patients can not properly express their complaints,such as psychosis, severe neurosis.
6. Taking NSIAD or alcohol abusers.
7. Allergic to penicillin or either drugs of the 6 antibiotic tested by susceptibility testing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Eradication rates | Three months
  To investigate the eradication rates of H.Pylori after individual quadruple therapy based on antibiotic susceptibility testing, CYP2C19 gene polymorphism, drug resistance gene sequencing and 16SrRNA sequencing.
Mutation site of drug resistance gene | Three months
  To discover the difference of mutation site in drug resistance gene between successful patients and refractory patients by second-generation sequencing.
The distribution and proportion of microflora in stomach | Three months
  To discover the distribution and proportion of microflora in stomach between successful patients and refractory patients of H. Pylori infection by 16SrRNA sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Youming Li, professor, Principal Investigator — First Affiliated Hospital of Zhejiang University